CLINICAL TRIAL: NCT00389441
Title: A Pivotal Phase 2 Study Of The Anti-Angiogenesis Agent AG-013736 In Patients With 131I-Refractory Metastatic Or Unresectable Locally-Advanced Thyroid Cancer
Brief Title: Study Of AG-013736 In Patients With 131I-Refractory Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: A4061027
Record Dates: First submitted 2006-10-16; First posted 2006-10-18 (Estimated); Results first posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-09

CONDITIONS: Thyroid Neoplasms
Keywords: VEGFR inhibitor; tyrosine kinase inhibitor; anti-angiogenic; carcinoma; papillary; follicular; medullary; anaplastic
MeSH Terms: conditions — Thyroid Neoplasms; Carcinoma | interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: AG-013736

INTERVENTIONS:
Drug: AG-013736 — AG-013736, tablets 5 mg BID , treatment will continue until tumor progression or toxicity

SUMMARY:
The primary purpose is to determine how effective AG-013736 is in shrinking thyroid cancer that is resistant to radioactive iodine

DETAILED DESCRIPTION:
Additional study details: assess safety and efficacy

ELIGIBILITY:
Inclusion Criteria:

* Radioiodine-refractory metastatic or unresectable locally-advanced thyroid cancer
* At least 1 measurable target lesion, as defined by RECIST

Exclusion Criteria:

* Thyroid lymphoma
* Previous treatment with anti-angiogenesis agents
* No myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, deep vein thrombosis or pulmonary embolism within 12 months prior.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2006-12; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (23):
- United States (8):
  - Pfizer Investigational Site, Orange, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Witchita, Kansas
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Buffalo, New York
- Canada (3):
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
- China (3):
  - Pfizer Investigational Site, Nanjing, Jiangsu
  - Pfizer Investigational Site, Beijing
  - Pfizer Investigational Site, Shanghai
- Pfizer Investigational Site, Prague, Czechia
- Pfizer Investigational Site, Vellore, Tamil Nadu, India
- Italy (2):
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Pisa
- Poland (2):
  - Pfizer Investigational Site, Gliwice
  - Pfizer Investigational Site, Warsaw
- Spain (2):
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Pamplona, Navarre
- Pfizer Investigational Site, Glasgow, United Kingdom

REFERENCES:
- [Derived] Locati LD, Licitra L, Agate L, Ou SH, Boucher A, Jarzab B, Qin S, Kane MA, Wirth LJ, Chen C, Kim S, Ingrosso A, Pithavala YK, Bycott P, Cohen EE. Treatment of advanced thyroid cancer with axitinib: Phase 2 study with pharmacokinetic/pharmacodynamic and quality-of-life assessments. Cancer. 2014 Sep 1;120(17):2694-703. doi: 10.1002/cncr.28766. Epub 2014 May 20. PMID 24844950
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4061027&StudyName=Study%20Of%20AG-013736%20In%20Patients%20%20With%20131I-Refractory%20thyroid%20cancer%20%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Axitinib: Axitinib (AG-013736) tablet 5 milligram (mg) orally twice daily continuously in 28-day cycles until tumor progression, unmanageable toxicity, or withdrawal of consent occurred. Dose was increased (to 7 mg or 10 mg twice daily) or decreased (to 3 mg or 2 mg twice daily) based on the tolerability.
Period: Overall Study
Arm/Group | Axitinib
Started | 52
Completed | 0
Not Completed | 52
Not completed — Adverse Event | 7
Not completed — Death | 4
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 4
Not completed — Physician Decision | 1
Not completed — Protocol Violation | 1
Not completed — Global deterioration of health status | 4
Not completed — Objective progression or relapse | 26
Not completed — Ongoing in study A4061008 (NCT00828919) | 2
Not completed — Clinical progression | 1

BASELINE CHARACTERISTICS:
Arm/Group | Axitinib
Number analyzed (Participants) | 52
Age Continuous [Mean (Standard Deviation); unit: years] | 57.6 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 28

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response (OR)
Description: Percentage of participants with OR based on assessment of confirmed complete response (CR) or confirmed partial response (PR) as per Response Evaluation Criteria in Solid Tumors (RECIST). CR: disappearance of all target/non-target lesions and no appearance of new lesions. PR: at least (>=)30 percent(%) decrease in sum of the longest dimensions (LDs) of the target lesions (taking as a reference the baseline sum), without progression of non-target lesions and no appearance of new lesions. Confirmed responses: those persist on repeat imaging study >=4 weeks after initial documentation of response.
Time Frame: Baseline until disease progression or initiation of antitumor therapy or death due to any cause, assessed every 8 weeks up to 28 days after last dose (follow-up)
Population: Intent-to-Treat (ITT) population included all participants who were enrolled in the study and received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Axitinib
Number analyzed (Participants) | 52
percentage of participants | 34.6 [22.0 to 49.1]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS: Time in weeks from the start of study treatment to first documentation of objective disease progression or to death due to any cause, whichever occurred first. PFS was calculated as (first event date minus the date of first dose of study treatment plus 1) divided by 7. Progression is defined using RECIST, as >=20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD since start of study and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions.
Time Frame: as for outcome 1
Population: ITT population included all participants who were enrolled in the study and received at least 1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Axitinib
Number analyzed (Participants) | 52
weeks | 70.14 [64.14 to 93.71]

3. Secondary Outcome: Duration of Response (DR)
Description: Time in weeks from the first documentation of objective tumor response to objective tumor progression or death due to any cause. Duration of tumor response was calculated as (the date of the first documentation of objective tumor progression or death due to any cause minus the date of the first CR or PR that was subsequently confirmed plus 1) divided by 7. DR was calculated for the subgroup of participants with a confirmed objective tumor response.
Time Frame: as for outcome 1
Population: Subgroup of participants from the ITT population, with a confirmed objective tumor response (CR or PR).
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Axitinib
Number analyzed (Participants) | 18
weeks | 74.71 [59.14 to 112.29]

4. Secondary Outcome: Overall Survival (OS)
Description: Time in weeks from the start of study treatment to date of death due to any cause. OS was calculated as (the death date minus the date of first dose of study medication plus 1) divided by 7. Death was determined from adverse event data (where outcome was death) or from follow-up contact data (where the participant current status was death).
Time Frame: Baseline to death due to any cause or at least 2 year after the first dose for the last participant
Population: ITT population included all participants who were enrolled in the study and received at least 1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Axitinib
Number analyzed (Participants) | 52
weeks | 118.43 [63.57 to 174.57]

5. Secondary Outcome: Change From Baseline in MD Anderson Symptom Assessment Inventory (MDASI) Symptom Severity Score
Description: Symptom severity score is comprised of average of 13 MDASI core items (pain, fatigue, nausea, disturbed sleep, distressed, shortness of breath, remembering things, lack of appetite, drowsy, dry mouth, sadness, vomiting, numbness or tingling). Participants were asked to rate severity of each symptom at their worst in last 24 hours; each item rated from 0 to 10, with 0 = symptom not present and 10 = as bad as you can imagine. Total average score range: 0 to 10. Lower scores indicated better outcome.
Time Frame: Baseline, Cycle 1 Day 15 (C1D15), C2D1, C2D15, thereafter D1 of each cycle up to 28 days after last dose (follow-up)
Population: ITT population included all participants who were enrolled in the study and received at least 1 dose of study treatment. Here 'N' (number of participants analyzed) signifies participants who were evaluable for this measure and 'n' signifies participants evaluable at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Axitinib
Number analyzed (Participants) | 49
units on a scale
  Baseline (n= 49) | 1.66 (1.301)
  Change at C1D15 (n= 40) | 0.18 (1.158)
  Change at C2D1 (n= 42) | 0.43 (1.274)
  Change at C2D15 (n= 37) | 0.52 (1.407)
  Change at C3D1 (n= 43) | 0.53 (1.602)
  Change at C4D1 (n= 39) | 0.58 (1.199)
  Change at C5D1 (n= 36) | 0.69 (1.550)
  Change at C6D1 (n= 36) | 0.53 (1.484)
  Change at C7D1 (n= 29) | 0.40 (1.344)
  Change at C8D1 (n= 28) | 0.44 (1.395)
  Change at C9D1 (n= 27) | 0.56 (1.516)
  Change at C10D1 (n= 25) | 0.59 (1.494)
  Change at C11D1 (n= 25) | 0.63 (1.669)
  Change at C12D1 (n= 24) | 0.59 (1.584)
  Change at C13D1 (n= 24) | 0.60 (1.281)
  Change at C14D1 (n= 24) | 0.59 (1.476)
  Change at C15D1 (n= 24) | 0.76 (1.654)
  Change at C16D1 (n= 23) | 0.81 (1.911)
  Change at C17D1 (n= 20) | 0.73 (1.816)
  Change at C18D1 (n= 20) | 0.60 (1.729)
  Change at C19D1 (n= 18) | 0.40 (1.201)
  Change at C20D1 (n= 16) | 0.50 (0.864)
  Change at C21D1 (n= 16) | 0.84 (1.094)
  Change at C22D1 (n= 15) | 0.61 (0.970)
  Change at C23D1 (n= 14) | 0.87 (1.086)
  Change at C24D1 (n= 11) | 1.05 (0.990)
  Change at C25D1 (n= 11) | 0.87 (1.016)
  Change at C26D1 (n= 9) | 1.15 (0.960)
  Change at C27D1 (n= 9) | 1.19 (1.244)
  Change at C28D1 (n= 10) | 0.95 (1.291)
  Change at C29D1 (n= 10) | 0.98 (1.080)
  Change at C30D1 (n= 10) | 1.03 (0.970)
  Change at C31D1 (n= 9) | 1.14 (1.100)
  Change at C32D1 (n= 9) | 1.44 (1.058)
  Change at C33D1 (n= 9) | 1.32 (1.233)
  Change at C34D1 (n= 8) | 1.54 (1.366)
  Change at C35D1 (n= 6) | 1.29 (1.233)
  Change at C36D1 (n= 6) | 1.27 (1.610)
  Change at C37D1 (n= 5) | 1.48 (1.347)
  Change at C38D1 (n= 5) | 1.27 (1.117)
  Change at C39D1 (n= 5) | 1.49 (1.288)
  Change at C40D1 (n= 5) | 1.47 (1.176)
  Change at C41D1 (n= 5) | 1.48 (1.267)
  Change at C42D1 (n= 5) | 1.59 (1.312)
  Change at C43D1 (n= 5) | 1.59 (1.259)
  Change at C44D1 (n= 5) | 1.42 (1.258)
  Change at C45D1 (n= 4) | 1.49 (1.349)
  Change at C46D1 (n= 4) | 1.73 (1.425)
  Change at C47D1 (n= 4) | 1.70 (1.543)
  Change at C48D1 (n= 3) | 1.90 (1.377)
  Change at C49D1 (n= 3) | 2.26 (1.554)
  Change at C50D1 (n= 3) | 2.38 (1.425)
  Change at C51D1 (n= 3) | 2.46 (1.533)
  Change at C52D1 (n= 1) | 3.38 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Change at C53D1 (n= 1) | 3.54 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Change at C54D1 (n= 1) | 3.00 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Change at C55D1 (n= 1) | 3.38 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Change at C56D1 (n= 1) | 3.15 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Change at C57D1 (n= 1) | 3.62 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Change at C58D1 (n= 1) | 3.23 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Change at C59D1 (n= 1) | 3.08 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Change at C60D1 (n= 1) | 3.85 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Change at C61D1 (n= 1) | 3.31 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Change at C62D1 (n= 1) | 3.46 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Change at follow-up (n= 12) | 0.37 (0.939)

6. Secondary Outcome: Change From Baseline in MD Anderson Symptom Assessment Inventory (MDASI) Symptom Interference Score
Description: Symptom interference score is comprised of average of 6 function items from MDASI core (general activity, mood, work, relations with others, walking, and enjoyment of life). Participants were asked to rate how much symptoms have interfered in last 24 hours; each item rated from 0 to 10, with 0 = did not interfere and 10 = interfered completely. Total average score range: 0 to 10. Lower scores indicated better outcome.
Time Frame: Baseline, Cycle 1 Day 15 (C1D15), C2D1, C2D15, thereafter D1 of each cycle up to 28 days after last dose (follow-up)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Axitinib
Number analyzed (Participants) | 48
units on a scale
  Baseline (n= 48) | 2.24 (2.193)
  Change at C1D15 (n= 40) | -0.05 (2.161)
  Change at C2D1 (n= 41) | 0.28 (2.763)
  Change at C2D15 (n= 36) | 0.67 (2.403)
  Change at C3D1 (n= 42) | 0.46 (2.669)
  Change at C4D1 (n= 37) | 0.47 (2.311)
  Change at C5D1 (n= 36) | 0.50 (2.377)
  Change at C6D1 (n= 36) | 0.65 (2.605)
  Change at C7D1 (n= 29) | 0.19 (2.386)
  Change at C8D1 (n= 28) | 0.22 (2.242)
  Change at C9D1 (n= 27) | 0.46 (2.450)
  Change at C10D1 (n= 25) | 0.35 (2.386)
  Change at C11D1 (n= 25) | 0.51 (2.784)
  Change at C12D1 (n= 23) | 0.32 (2.593)
  Change at C13D1 (n= 24) | 0.42 (2.346)
  Change at C14D1 (n= 24) | 0.42 (2.624)
  Change at C15D1 (n= 24) | 0.69 (2.902)
  Change at C16D1 (n= 23) | 0.73 (3.179)
  Change at C17D1 (n= 20) | 0.26 (2.920)
  Change at C18D1 (n= 20) | 0.35 (2.638)
  Change at C19D1 (n= 18) | -0.18 (2.497)
  Change at C20D1 (n= 15) | 0.30 (2.124)
  Change at C21D1 (n= 15) | 0.50 (1.954)
  Change at C22D1 (n= 14) | 0.32 (1.979)
  Change at C23D1 (n= 14) | 0.95 (1.615)
  Change at C24D1 (n= 11) | 0.77 (1.844)
  Change at C25D1 (n= 11) | 0.65 (1.699)
  Change at C26D1 (n= 9) | 1.04 (1.681)
  Change at C27D1 (n= 9) | 0.81 (2.463)
  Change at C28D1 (n= 28) | 0.67 (1.956)
  Change at C29D1 (n= 29) | 0.88 (1.926)
  Change at C30D1 (n= 30) | 1.03 (1.846)
  Change at C31D1 (n= 9) | 1.19 (1.910)
  Change at C32D1 (n= 9) | 1.52 (1.870)
  Change at C33D1 (n= 9) | 1.07 (1.972)
  Change at C34D1 (n= 8) | 1.81 (1.846)
  Change at C35D1 (n= 6) | 1.17 (1.517)
  Change at C36D1 (n= 6) | 0.97 (1.572)
  Change at C37D1 (n= 5) | 1.40 (1.782)
  Change at C38D1 (n= 5) | 1.23 (1.521)
  Change at C39D1 (n= 5) | 1.50 (1.453)
  Change at C40D1 (n= 5) | 1.83 (1.889)
  Change at C41D1 (n= 5) | 1.53 (1.746)
  Change at C42D1 (n= 5) | 1.67 (1.637)
  Change at C43D1 (n= 5) | 1.31 (1.267)
  Change at C44D1 (n= 5) | 1.34 (1.345)
  Change at C45D1 (n= 4) | 1.50 (1.694)
  Change at C46D1 (n= 4) | 2.17 (2.113)
  Change at C47D1 (n= 4) | 1.63 (1.950)
  Change at C48D1 (n= 3) | 2.00 (1.041)
  Change at C49D1 (n= 3) | 2.56 (1.798)
  Change at C50D1 (n= 3) | 0.22 (1.206)
  Change at C51D1 (n= 3) | 2.44 (1.251)
  Change at C52D1 (n= 1) | 3.33 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Change at C53D1 (n= 1) | 3.33 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Change at C54D1 (n= 1) | 3.33 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Change at C55D1 (n= 1) | 3.50 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Change at C56D1 (n= 1) | 3.50 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Change at C57D1 (n= 1) | 4.50 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Change at C58D1 (n= 1) | 3.67 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Change at C59D1 (n= 1) | 3.33 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Change at C60D1 (n= 1) | 4.83 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Change at C61D1 (n= 1) | 3.33 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Change at C62D1 (n= 1) | 4.00 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Change at follow-up (n= 12) | 0.32 (2.396)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Axitinib
Serious Adverse Events (participants affected / at risk) | 22/52
Other Adverse Events (participants affected / at risk) | 52/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib (N=52)
Cardiac failure congestive (Cardiac disorders) | 1
Hypertensive heart disease (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Disease progression (General disorders) | 2
Fatigue (General disorders) | 3
Hypersensitivity (Immune system disorders) | 1
Appendicitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Weight decreased (Investigations) | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral ischaemia (Nervous system disorders) | 1
Monoplegia (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Arteriosclerosis (Vascular disorders) | 1
Jugular vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib (N=52)
Anaemia (Blood and lymphatic system disorders) | 3
Leukocytosis (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Paratracheal lymphadenopathy (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Atrial thrombosis (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Phimosis (Congenital, familial and genetic disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Hypoacusis (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Hyperparathyroidism (Endocrine disorders) | 1
Hyperparathyroidism secondary (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 3
Cataract (Eye disorders) | 1
Conjunctival haemorrhage (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 2
Diplopia (Eye disorders) | 1
Eye swelling (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 1
Orbital oedema (Eye disorders) | 1
Periorbital oedema (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Vitreous floaters (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 5
Abdominal pain upper (Gastrointestinal disorders) | 8
Barrett's oesophagus (Gastrointestinal disorders) | 1
Chapped lips (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Colonic polyp (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 31
Dry mouth (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Gingival bleeding (Gastrointestinal disorders) | 2
Glossodynia (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 3
Haemorrhoids (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 14
Odynophagia (Gastrointestinal disorders) | 2
Oral pain (Gastrointestinal disorders) | 1
Proctitis (Gastrointestinal disorders) | 2
Rectal haemorrhage (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 6
Tongue ulceration (Gastrointestinal disorders) | 2
Toothache (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 7
Asthenia (General disorders) | 4
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 3
Facial pain (General disorders) | 1
Fatigue (General disorders) | 23
Feeling cold (General disorders) | 2
Gait disturbance (General disorders) | 2
Mucosal inflammation (General disorders) | 10
Oedema peripheral (General disorders) | 4
Pain (General disorders) | 3
Pyrexia (General disorders) | 4
Cholecystitis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 2
Anal abscess (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Candidiasis (Infections and infestations) | 1
Dermatitis infected (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Herpes simplex ophthalmic (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Influenza (Infections and infestations) | 5
Laryngitis (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 4
Otitis externa (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Parotitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 3
Procedural pain (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase (Investigations) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Blood cholesterol increased (Investigations) | 1
Blood creatinine increased (Investigations) | 3
Blood lactate dehydrogenase increased (Investigations) | 2
Blood phosphorus increased (Investigations) | 1
Blood pressure decreased (Investigations) | 1
Blood pressure diastolic increased (Investigations) | 1
Blood pressure increased (Investigations) | 4
Blood thyroid stimulating hormone decreased (Investigations) | 1
Blood thyroid stimulating hormone increased (Investigations) | 3
Crystal urine present (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Haematocrit increased (Investigations) | 1
Haemoglobin increased (Investigations) | 5
Platelet count decreased (Investigations) | 1
Protein urine present (Investigations) | 2
Thyroglobulin increased (Investigations) | 1
Thyroxine increased (Investigations) | 2
Weight decreased (Investigations) | 18
Decreased appetite (Metabolism and nutrition disorders) | 19
Dehydration (Metabolism and nutrition disorders) | 1
Gout (Metabolism and nutrition disorders) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 9
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Mastication disorder (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1
Lipofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ataxia (Nervous system disorders) | 1
Burning sensation (Nervous system disorders) | 1
Disturbance in attention (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 4
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 10
Hypoaesthesia (Nervous system disorders) | 2
Lethargy (Nervous system disorders) | 1
Motor dysfunction (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 4
Paraesthesia (Nervous system disorders) | 7
Somnolence (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 1
Thrombotic cerebral infarction (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 5
Insomnia (Psychiatric disorders) | 5
Mood altered (Psychiatric disorders) | 1
Sleep disorder (Psychiatric disorders) | 2
Dysuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 2
Pollakiuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 6
Urinary retention (Renal and urinary disorders) | 1
Urinary tract pain (Renal and urinary disorders) | 2
Amenorrhoea (Reproductive system and breast disorders) | 1
Dyspareunia (Reproductive system and breast disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 2
Menstrual disorder (Reproductive system and breast disorders) | 2
Pelvic pain (Reproductive system and breast disorders) | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 11
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 6
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 7
Dermal cyst (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 5
Eczema (Skin and subcutaneous tissue disorders) | 3
Erythema (Skin and subcutaneous tissue disorders) | 1
Hair colour changes (Skin and subcutaneous tissue disorders) | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 1
Nail pigmentation (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 6
Petechiae (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 8
Skin disorder (Skin and subcutaneous tissue disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 1
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 1
Skin swelling (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Mole excision (Surgical and medical procedures) | 1
Hypertension (Vascular disorders) | 28
Hypertensive crisis (Vascular disorders) | 1
Peripheral artery thrombosis (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.